CLINICAL TRIAL: NCT05189678
Title: Correlation Between Modified Weakness Index and Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Surgery: a Single-center Prospective Observational Cohort Study
Brief Title: Correlation Between Modified Weakness Index and Postoperative Delirium in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: Frailty
Record Dates: First submitted 2021-12-13; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Frailty
Keywords: Frailty POD
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- frailty group: Modified Frailty index score greater than or equal to 0.21
  Interventions: Other: No intervention
- non-frailty group: Modified Frailty index score is less than 0.21
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
1. To study whether there is a correlation between weakness and postoperative delusions in elderly non-cardiac surgery patients
2. Can the improved debilitating index predict the delusion after non-cardiac surgery
3. Which of the debilitating index are independent risk factors associated with postoperative delusions

DETAILED DESCRIPTION:
Early identification of frailty patients is of great clinical significance for preoperative decision making and prognosis assessment. To date, the incidence of postoperative delirium in elderly patients undergoing noncardiac surgery has not been assessed. This study aimed to investigate the relationship between preoperative frailty assessment and the incidence of postoperative delirium after noncardiac surgery.

1. To study whether there is a correlation between weakness and postoperative delusions in elderly non-cardiac surgery patients
2. Can the improved debilitating index predict the delusion after non-cardiac surgery
3. Which of the debilitating index are independent risk factors associated with postoperative delusions

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years old;
2. ASA: Grade Ⅰ～Ⅳ;
3. Signed informed consent；
4. Scheduled non-cardiac surgery.

Exclusion Criteria:

1. Refuse to participate;
2. Expected length of stay <3 days;
3. The same patient can only be included once, regardless of whether the reason for the second operation is related to the first cause;
4. Emergency surgery patients;
5. Inability to communicate due to illiteracy, language impairment, severe hearing or visual impairment;
6. Central nervous system diseases, including various types of dementia and depression
7. Severe renal insufficiency (requiring dialysis treatment);
8. Severe liver dysfunction (Child-Pugh score ≥10);
9. Patients who have participated in other relevant clinical studies within 3 months MMSE examination has confirmed the existence of cognitive dysfunction: illiteracy ≤17 points, primary school degree ≤20 points, middle school degree (including technical secondary school) ≤22 points, university degree (including junior college) ≤23 points

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 70 years undergoing non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium | Twice a day from day 1 to 3 after surgery (8:00-10:00 am and 18:00-20:00 PM).
  Incidence of postoperative delirium after noncardiac surgery.Postoperative delirium usually occurs between 24 hours and 72 hours after surgery, and this study will conduct follow-up assessments at six postoperative time points (once in the morning and afternoon on days 1 to 3 after surgery, 8:00 a.m.-10:00 a.m., 18:00-20:00 pm), as long as there was one time point to assess postoperative delirium, the patient was judged to have developed postoperative delirium.

SECONDARY OUTCOMES:
Incidence of 30-day readmission to hospital | Within 30 days after surgery
  Incidence of 30-day readmission to hospital
complications | Within 30 days after surgery
  Patients were followed up 30 days later for complications

CONTACTS AND LOCATIONS:
Overall Officials: Yuelan Wang, PhD, Principal Investigator — Shandong First Medical University
Locations (1):
- Yongtao Sun, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kulason K, Nouchi R, Hoshikawa Y, Noda M, Okada Y, Kawashima R. Indication of Cognitive Change and Associated Risk Factor after Thoracic Surgery in the Elderly: A Pilot Study. Front Aging Neurosci. 2017 Dec 5;9:396. doi: 10.3389/fnagi.2017.00396. eCollection 2017. PMID 29259553
- [Result] Woo J, Yu R, Wong M, Yeung F, Wong M, Lum C. Frailty Screening in the Community Using the FRAIL Scale. J Am Med Dir Assoc. 2015 May 1;16(5):412-9. doi: 10.1016/j.jamda.2015.01.087. Epub 2015 Feb 24. PMID 25732832
- [Result] Gleason LJ, Benton EA, Alvarez-Nebreda ML, Weaver MJ, Harris MB, Javedan H. FRAIL Questionnaire Screening Tool and Short-Term Outcomes in Geriatric Fracture Patients. J Am Med Dir Assoc. 2017 Dec 1;18(12):1082-1086. doi: 10.1016/j.jamda.2017.07.005. Epub 2017 Aug 31. PMID 28866353
- [Derived] Zhang M, Gao X, Liu M, Gao Z, Guo Y, Chen L, Liu Y, Zhang X, Huang L, Tong M, Zou T, Sun Y. Correlation of preoperative frailty with postoperative delirium and 1-year mortality in Chinese geriatric patients undergoing non-cardiac surgery: a prospective observational cohort study. Int J Surg. 2025 Jan 1;111(1):1576-1579. doi: 10.1097/JS9.0000000000002042. No abstract available. PMID 39166961
- [Derived] Zhang M, Gao X, Liu M, Gao Z, Sun X, Huang L, Zou T, Guo Y, Chen L, Liu Y, Zhang X, Feng H, Wang Y, Sun Y. Correlation of preoperative frailty with postoperative delirium and one-year mortality in Chinese geriatric patients undergoing noncardiac surgery: Study protocol for a prospective observational cohort study. PLoS One. 2024 Mar 6;19(3):e0295500. doi: 10.1371/journal.pone.0295500. eCollection 2024. PMID 38446754